CLINICAL TRIAL: NCT07283822
Title: A Phase II Trial of JAK Inhibitor Added to Immunotherapy for Treatment of Relapsed/Refractory T-cell Lymphoma and 9p Amplified Lymphomas
Brief Title: Amping up With PemJAK
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Seda S. Tolu (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor-Investigator, Seda S. Tolu, Assistant Professor of Medicine, Columbia University
Organization: Columbia University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AAAV7563
Record Dates: First submitted 2025-12-06; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Non-Hodgkin Lymphoma; Hodgkin Disease Lymphoma; Non-Hodgkin Lymphoma Refractory/ Relapsed; Hodgkin Disease Recurrent; Gray Zone Lymphoma; Peripheral T-cell Lymphoma; Cutaneous T-Cell Lymphomas; Primary Mediastinal B Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, T-Cell, Peripheral; Lymphoma, T-Cell, Cutaneous | interventions — ruxolitinib; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib (Experimental): Ruxolitinib 20mg PO twice daily will be continued until 12 months, disease progression, or development of intolerable side effects (whichever occurs first).
  Interventions: Drug: Ruxolitinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Ruxolitinib — Patients will receive the study drug ruxolitinib for as long as the disease responds, for up to a maximum of one year (or 17 cycles). After study treatment with ruxolitinib is finished, the study doctor will continue to watch for side effects and follow the condition for one year. If any side effects are experienced, the study doctor will follow up until resolution or stabilization of the side effect.
Drug: Pembrolizumab — Pembrolizumab immunotherapy will be administered intravenously at 200 mg once every 21 days. Subjects will receive pembrolizumab for as long as the disease responds, up to a maximum of one year (or 17 cycles). Each cycle is 21 days long.

SUMMARY:
The purpose of this study is to understand and determine if ruxolitinib added to pembrolizumab is safe and effective for the treatment of relapsed or refractory Hodgkin and non-Hodgkin lymphomas.

DETAILED DESCRIPTION:
This study includes peripheral T-cell lymphoma (PTCL), cutaneous T-cell lymphomas (CTCL), and other lymphomas (Hodgkin Lymphoma [HL], Gray Zone Lymphomas [GZL], and Primary Mediastinal B-cell Lymphoma [PMBCL]) that has become resistant to commonly available chemotherapy (refractory), or it has re-occurred after treatment (relapsed). For PTCL participants, the main goal is to see how many achieve complete remission (no signs of cancer). For CTCL participants, the focus is on the overall response rate, meaning how many show improvement. This study is also open to patients with Hodgkin Lymphoma (HL), Gray Zone Lymphoma (GZL), and Primary Mediastinal B-cell Lymphoma (PMBCL), to understand if ruxolitinib can work in a disease that shares similar characteristics. It is important to note that ruxolitinib is an investigational drug and is not FDA approved for these lymphomas, but has shown to be effective in combination with immunotherapy in clinical trials. In addition, pembrolizumab is only FDA approved for HL and PMBCL - however is commonly used in PTCL, CTCL, and GZL in the relapsed setting as treatment options are limited and prior trials with pembrolizumab has shown effectiveness in treating these lymphomas.

ELIGIBILITY:
Inclusion Criteria:

* (1) Histologically confirmed relapsed/refractory HL, PMBCL, GZL, and TCL including the below subtypes:

  * Arm 1: PTCL

    * Nodal PTCL Peripheral T-cell Lymphoma- Not Otherwise Specified (PTCL-NOS)
    * Anaplastic Large Cell Lymphoma (ALCL) T-follicular Helper Lymphomas (TFH) and its subtypes including angioimmunoblastic T-cell Lymphoma (AITL)
    * Extranodal NK/T-cell lymphoma
    * Subcutaneous Panniculitis T-Cell Lymphoma
  * Arm 2: CTCL

    * Mycosis Fungoides
    * Sezary Syndrome
  * Arm 3: exploratory cohort

    * Classic HL
    * PMBCL
    * GZL
* (2) All patients must have received at least one-line systemic therapy.

  * Patients with systemic ALCL must have received prior CD30-directed therapy.
  * Other PTCL subtypes that express CD30 (>10%), must have received prior CD30-directed therapy.
  * Special Consideration for CTCL in Arm 2:

    * Systemic therapies including bexarotene (targretin) are permissible up to 2 weeks prior to enrollment.
    * Skin directed therapies including light therapy/phototherapy, extracorporeal photopheresis (ECP), topical steroids, or mechlorethamine (valchlor) gel are NOT considered a systemic line of therapy when given alone.
    * Treatment with radiation, phototherapy, histone deacetylase inhibitor, retinoids, interferons, therapeutic doses of systemic corticosteroids, or denileukin diftitox (18 µg/kg/day) up to 2 weeks prior to enrollment is allowed.
    * Treatment with alemutuzumab up to 8 weeks prior to enrollment is permissible.
* (3) Patients must not have had chemotherapy or immunotherapy within 2 weeks prior to entering the study and must have recovered from adverse events (to grade 1 or less)
* (4) Anti PD-1/PDL-1is permissible up to two weeks prior to enrollment.
* (5) Age ≥ 18
* (6) Participants must have measurable disease, as defined in the protocol

  * Patients must have a PET-CT scan performed within ≤4 weeks.
  * Contrast enhanced CT scan or MRI of the neck, chest, abdomen, pelvis is permissible, however; PET is preferred.
* (7) Patients cannot have active central nervous system (CNS) disease. Patients that have been treated and asymptomatic are allowed on study.
* (8) All participants must be screened for chronic hepatitis B virus (HBV) with hepatitis B viral load and serologies (core antibody, surface antigen, and surface antibody) within 30 days prior to enrollment.

  * Patients with positive Hep B core will need to be on HBV prophylaxis
  * Patients with positive Hep B core will need to be on HBV prophylaxis.
* (9) Participants with a history of hepatitis C virus (HCV) infection must have been treated and cured. If actively on treatment, HCV viral load mut be undetectable 30 days prior to enrollment.
* (10) Participants with known human immunodeficiency virus (HIV)-infection are eligible providing they are on effective anti-retroviral therapy and have undetectable viral load at their most recent viral load test (must be within 26 weeks prior to enrollment).
* (11) Organ function as assessed by laboratory testing and Eastern Cooperate Oncology Group (ECOG) performance status 0-2 and or a Karnofsky performance score of equal or greater to 50 (see Section 20.1.1, Appendix A) for receipt of ruxolitinib and pembrolizumab.

  * Absolute Neutrophil Count ≥ 1000/μL (not growth factor independent)
  * Platelets ≥ 70,000/μL (or ≥50,000/mm3 if known bone marrow involvement with dose modifications allowed. See protocol for specific instructions for dose modifications).
  * Baseline hemoglobin level ≥ 8 g/dL (irrespective of bone marrow involvement).
  * Calculated creatinine clearance ≥ 30 ml/min using the Cockcroft-Gault formula
  * Bilirubin ≤ 2 x upper limit of normal (ULN)
  * Aspartate aminotransferase (AST) ≤ 2.5 × ULN
  * Alanine aminotransferase (ALT) ≤ 2.5 × ULN
* (12) Ability to understand and the willingness to sign a written informed consent document.
* (13) Patients with prior history of deep vein thrombosis (DVT) that has been treated or actively requiring anticoagulation are permitted to enroll.
* (14) Due to the potential teratogenic effects, women of childbearing age must have a documented negative serum β-hCG measured within 2 weeks of starting treatment. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician and Incyte immediately (see protocol). Additionally, both women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence).

Contraception should continue for 6 months after you stop taking study drug. Similarly, women must agree to not breastfeed during the entirety of the study period.

Exclusion Criteria:

* 1) Diagnosis of Adult T-Cell Leukemia/Lymphoma (ATLL)
* 2) History of autoimmune disease that requires systemic treatment.
* 3) Has a diagnosis of immunodeficiency or receiving immunosuppressive therapy within 7 days prior to the first dose of study drug.
* 4) Actively chronic systemic steroids therapy (in dosing exceeding 10mg daily of prednisone or its drug equivalent).

  o Patients must be off steroid therapy exceeding 10mg or greater of prednisone (or its equivalent) at the start of therapy.
* 5) Patients with HL and PMBCL patients must not be eligible and agreeable to autologous stem cell transplant.

  o Patients with PMBCL must not be eligible and agreeable to CAR-T.
* 6) Allowed to have disease progression after or refractory to autologous bone marrow transplant.
* 7) Progression after allogeneic stem cell transplantation (SCT) can be determined on a case-by-case basis after discussion with the primary investigator.
* 8) History of solid organ transplant requiring active immunosuppression for which treatment with immunotherapy would be contraindicated.
* 9) Active TB (Tuberculosis Bacillus) at time screening. Prior cases of adequately treated TB are permissible.
* 10) Has severe hypersensitivity (≥ Grade 3) to pembrolizumab and/or any of its excipients.
* 11) Has severe hypersensitivity (≥ Grade 3) to ruxolitinib and/or any of its excipients.

Patients with G1 and G2 hypersensitivity remain eligible.

* 12) Inability to swallow or take medications by mouth
* 13) Is pregnant or breastfeeding or expected to conceive children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of trial treatment.
* 14) History of concurrent and active malignancy for which he or she is currently receiving directed therapy for.
* 15) History of major adverse cardiac events such as myocardial infraction or stroke within 6 months of enrollment. Cardiovascular events within 6 months such as pulmonary embolism and deep vein thrombosis is permissible if on therapeutic treatment.
* 16) Subjects with active, systemic, and uncontrolled bacterial, viral, or fungal infections at the time of screening will be excluded from study participation.

Exceptions include:

Infections that have been appropriately treated, with evidence of clinical resolution and return to baseline organ function within 14 days prior to study entry.

* Localized, non-systemic infections (e.g., uncomplicated urinary tract infections or cellulitis) that are being actively managed and are not associated with systemic symptoms.
* Please see section protocol for eligibility requirements specifically for HCV, HBV, HIV and Tuberculosis infections at time of screening.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2025-12-03 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) rate | 24 months from the start of study treatment
  For Arm 1, in patients with Peripheral T-cell Lymphoma (PTCL), the primary objective will be complete response (CR) rate.
Overall response rate (ORR) | 24 months from the start of study treatment
  For Arm 2, in patients with Cutaneous T-cell Lymphoma (CTCL), the primary objective will be overall response rate (ORR)

CONTACTS AND LOCATIONS:
Overall Officials: Seda Tolu, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States